CLINICAL TRIAL: NCT05697536
Title: Comparison of Pilates and Aerobic Exercises on Pain, Anxiety and Quality of Life in Premenstrual Syndrome
Brief Title: Comparison of Pilates and Aerobic Exercises on Pain, Anxiety and QOL in PMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Adeela Arif
Record Dates: First submitted 2023-01-04; First posted 2023-01-26 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Premenstrual Syndrome
MeSH Terms: conditions — Premenstrual Syndrome | interventions — Exercise Movement Techniques; Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pilates training (Experimental): Group A will receive Pilates training. The treatment will be given with the frequency of 3 times per week for 8 weeks. Treatment sessions will be of 45 minutes with short resting intervals.
  Interventions: Other: Pilates training
- Aerobic exercise (Experimental): Group B will receive aerobic exercise plan. The frequency of treatment will be as same as that of Pilates exercise program i.e. 3 times a week for 8 weeks. Treatment sessions will be of 45 minutes with short resting intervals.
  Interventions: Other: Aerobic Exercise

INTERVENTIONS:
Other: Pilates training — It consists of patients who will receive pilates exercise training sessions 3 times per week for 8 weeks. Every session will be of 45 minutes. Exercise programs follow the basic principles of pilates method but particularly movements with low and medium difficulty levels will be chosen to adapt the program to the physical capacity of the patients.
  Protocol will be compromise of 9 modules: postural education, search for neutral position, sitting exercise, antalgic exercise, stretching exercises, proprioceptively improvement exercises and breathing exercises.
  Arms: Pilates training
Other: Aerobic Exercise — It consists of patients who will receive aerobic exercise sessions 3 times per week for 8 weeks. Every session will be of 45 minutes.
  It will include warm up phase, active phase and
  Arms: Aerobic exercise

SUMMARY:
The significance of this study is that it may improve the premenstrual symptoms like pain and anxiety in females with premenstrual syndrome and improve their quality of life. This study may add to the growing body of knowledge that if these two techniques yield comparable outcomes and if one technique is superior to the other, which should be the alternative choice of therapy. Therefore, the study will be done to compare the effects of Pilate exercises and aerobic exercises on pain, anxiety and quality of life in females with premenstrual syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Unmarried
* Age between 18-30 years
* Patients with at least 5 of 11 symptoms on premenstrual syndrome questionnaire

Exclusion Criteria:

* Patients suffering from Any Disability.
* Patients suffering from diabetes or hypertension or any other Chronic Illness.
* Spine fracture or history of Any Previous Surgery.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 26 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2023-02-25 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | 8th week
  The Numerical pain rating scale is the most commonly used pain scale in the health care.
  This scale is used on subjects of age more than 9. By using this scale ask the participant to rate their pain orally by giving the numbers from 0-10. 0 means no pain and 10 worst pain.
Anxiety | 8th week
  DASS-21 is a self reported questionnaire which is used to assess the severity of range of symptoms like depression, anxiety and stress. It is not only used to measure the severity of symptoms but can also be used to assess the subject's response to treatment. Less the scores mean less anxiety and more the score means severe anxiety.
WHO quality of life questionnaire | 8th week
  WHO inventiveness to develop a quality of life assessment arises from a requirement for a genuinely international measure of quality of life and a commitment to the continued promotion of an holistic approach to health and health care. Its developmental process consisted of several stages.

CONTACTS AND LOCATIONS:
Overall Officials: Adeela Arif, Mphil, Principal Investigator — Riphah International University
Locations (1):
- Riphah International university, Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dickerson LM, Mazyck PJ, Hunter MH. Premenstrual syndrome. Am Fam Physician. 2003 Apr 15;67(8):1743-52. PMID 12725453
- [Background] Samadi Z, Taghian F, Valiani M. The effects of 8 weeks of regular aerobic exercise on the symptoms of premenstrual syndrome in non-athlete girls. Iran J Nurs Midwifery Res. 2013 Jan;18(1):14-9. PMID 23983722
- [Background] Citil ET, Kaya N. Effect of pilates exercises on premenstrual syndrome symptoms: a quasi-experimental study. Complement Ther Med. 2021 Mar;57:102623. doi: 10.1016/j.ctim.2020.102623. Epub 2020 Nov 24. PMID 33246104
- [Background] Roh SY. Effect of a 16-week Pilates exercise program on the ego resiliency and depression in elderly women. J Exerc Rehabil. 2016 Oct 31;12(5):494-498. doi: 10.12965/jer.1632704.352. eCollection 2016 Oct. PMID 27807531